CLINICAL TRIAL: NCT03739983
Title: Alterations in the Vaginal Microenvironment Using a Non-pharmacological Intervention for Breast Cancer Patients Treated With Aromatase Inhibitors
Brief Title: Alterations in the Vaginal Microenvironment Using a Non-pharmacological Intervention
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual as a result of COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW17032; 2018-0633 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH/OBSTET & GYNEC/GYNEC ONC (Other: UW Madison); NCI-2018-02729 (Registry Identifier: NCI Trial ID); Protocol Version 10/3/2019 (Other: UW Madison)
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-08

CONDITIONS: Adherence, Medication
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Prospective Simon two-stage study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VRP Therapy (Experimental): All subjects on this study will receive the Vaginal Renewal Program intervention. Enrolled subjects will receive inperson instruction on how to perform the VRP. Subjects will be encouraged to use the device for 3-4 days per week for 5 minutes at a time.
  Interventions: Device: Vaginal Renewal Program

INTERVENTIONS:
Device: Vaginal Renewal Program — Therapeutic vibrating wand.
  Other Names: FeMani Vibrating Massage Wand

SUMMARY:
Breast cancer patients commonly take medications to reduce the risk of recurrence, including aromatase inhibitors (AIs). AIs can cause significant side effects that reduce patient adherence. Early discontinuation of AI therapy results in an increased risk of cancer recurrence and increased risk of breast cancer-related death. Common side effects include vaginal dryness and vulvovaginal atrophy leading to worsening sexual function. To increase AI adherence, the investigators will study a non-pharmaceutical Vaginal Renewal Program (VRP) aimed at stimulating nitric oxide production to consequently increase vaginal lubrication, and improve the symptoms of vulvovaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Have completed active primary treatment

  * defined as surgery chemotherapy and/or radiation for the treatment of breast cancer
  * Does not include immunotherapy or other targeted therapies such as trastuzumab, CDK 4/6 or mTOR inhibitors
* Have been receiving AIs for at least 6 months prior to enrollment
* Plan to continue AIs for an additional 3 months
* Amenorrhea for at least 12 months at enrollment
* Participants must be able to read and write in English
* Participants must have < 2% superficial vaginal cells on cytologic evaluation

Exclusion Criteria:

* Pre-existing hypertonic pelvic floor dysfunction identified in the medical record
* Unresolved or recurrent vaginismus identified in the medical record
* Aversion to touching one's own body, including genitals, or using vibration therapy on the genitals
* Currently receiving estrogen therapy, including topical and/or systemic estrogens
* Have received estrogen therapy within 6 months of study enrollment, including topical and/or systemic estrogens
* Any surgical procedure to the vagina or vulva, excluding office biopsies, within the previous 12 months
* Receipt of pelvic or vaginal or vulvar radiation therapy within the 12 months prior to enrollment or if the subject is anticipated to receive radiation targeted to any of these 3 locations within 6 months following enrollment
* Any use of the VRP off study within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Spencer, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited with the help of the University of Wisconsin Carbone Cancer Center in November and December 2019. Recruitment was suspended in March 2020 due to the COVID-19 pandemic.
Period: Overall Study
Arm/Group | VRP Therapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VRP Therapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Superficial Vaginal Cells
Description: The investigators expect the percentage of superficial vaginal cells to be greater at the post-intervention time point when compared to the pre-intervention time point. If the percentage of superficial vaginal cells is ≥ 4% following the intervention, then the response will be considered positive.
Time Frame: up to 12 weeks
Population: End of study samples unavailable, decision was made not to analyze primary outcome as it was not powered to produce meaningful results.
Groups:
- VRP Therapy: All subjects on this study will receive the Vaginal Renewal Program (VRP) intervention. Enrolled subjects will receive inperson instruction on how to perform the VRP. Subjects will be encouraged to use the device for 3-4 days per week for 5 minutes at a time.
Arm/Group | VRP Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Vaginal pH
Description: Changes in the vaginal pH will be analyzed to determine the extent to which the changes correlate with changes in the primary outcome and with patient reported outcomes. Given the longitudinal nature of the study, linear and generalized linear mixed effects models will be fit to the data gathered. The restricted maximum likelihood (REML) criterion will be used and 95% semi-parametrically bootstrapped confidence intervals will be obtained for all parameters. All statistical analyses will be conducted using R (R Core Team 2014).
Time Frame: up to 12 weeks
Population: No data to analyze.
Arm/Group | VRP Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Patient Reported Outcomes: Number of Subjects With Improved Anxiety
Description: Number of subjects with improved anxiety outcomes per over baseline. The PROMIS (Patient Reported Outcomes Measurement Information System) Emotional Distress - Anxiety scale measures patient perceived changes in anxiety and includes 8 questions that they answer about their emotional state in the past 7 days. Descriptive answers are scored from 1 (never) to 5 (always). The total possible range of scores is from 8-40, with higher scores indicating a worse outcome.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VRP Therapy
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Patient Reported Outcomes: Number of Subjects With Improved Depression
Description: Number of subjects with improved depression outcomes over baseline. The PROMIS (Patient Reported Outcomes Measurement Information System) Emotional Distress - Depression scale measures patient perceived changes in depression and includes 8 questions that they answer about their emotional state in the past 7 days. Descriptive answers are scored from 1 (never) to 5 (always). The total possible range of scores is from 8-40, with higher scores indicating a worse outcome.
Time Frame: up to 12 weeks
Population: only 1 participant completed this survey
Measure: Count of Participants; unit: Participants
Arm/Group | VRP Therapy
Number analyzed (Participants) | 1
Participants | 0

5. Secondary Outcome: Patient Reported Outcomes: Number of Subjects With Improved Sexual Function Outcomes
Description: Number of subjects with improved sexual function outcomes over baseline. The PROMIS (Patient Reported Outcomes Measurement Information System) Sexual Function Profile scale measures patient perceived changes in sexual function and includes 10 questions that they answer about their functional state. Descriptive answers include 'Not at all', 'A little bit', 'Somewhat', 'Quite a bit', or 'Very', and will be summarized with descriptive statistics.
Time Frame: up to 12 weeks
Population: Incomplete data, unable to evaluate.
Arm/Group | VRP Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Patient Reported Outcomes: Number of Subjects With Improved Global Health
Description: Number of subjects with improved global health over baseline. The PROMIS (Patient Reported Outcomes Measurement Information System) Global Health scale measures patient perceived changes in health and includes 10 questions that they answer about their perceived health in the past 7 days. Higher scores indicate a higher perceived level of overall health.
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VRP Therapy
Number analyzed (Participants) | 2
Participants | 0

7. Secondary Outcome: Patient Reported Outcomes: Number of Subjects With Improved Sex Life
Description: Number of subjects with improved sex life over baseline. The PROMIS (Patient Reported Outcomes Measurement Information System) Global Satisfaction with Sex Life scale measures patient perceived changes in the satisfaction of their sex life and includes 7 questions that they answer about their perceived state. Descriptive answers include 'Not at all', 'A little bit', 'Somewhat', 'Quite a bit', or 'Very', and will be summarized with descriptive statistics.
Time Frame: up to 12 weeks
Population: Incomplete data, unable to evaluate.
Arm/Group | VRP Therapy
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Adherence to AI Therapy
Description: Adherence to AI therapy will be determined using patient-reported logs.
Time Frame: up to 12 weeks
Population: No data to analyze
Arm/Group | VRP Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | VRP Therapy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRP Therapy (N=2)
Irritation (Reproductive system and breast disorders) | 1 (1)
Vulvar Stinging (Reproductive system and breast disorders) | 1 (1)
Perineal Chaffing (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early with 2 participants due to the COVID-19 pandemic. It is not powered for meaningful results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03739983/Prot_SAP_000.pdf